CLINICAL TRIAL: NCT01499017
Title: A Phase 1, Randomized, Double Blind, Sponsor Open, Placebo-Controlled, Single Dose Escalating Study To Assess The Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Of PF-06291874 After Administration Under Fasted And Fed Conditions In Healthy Adult Subjects
Brief Title: A Single Dose Study Of PF-06291874 In Healthy Adult Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: B4801001
Record Dates: First submitted 2011-11-14; First posted 2011-12-26 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: Single Ascending Dose Study in healthy subjects
MeSH Terms: interventions — PF-06291874

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Experimental): Each subjects in Cohort A will receive 3 single doses of PF-06291874 and 1 placebo dose in random order in Periods 1-4.
  Interventions: Drug: PF-06291874 or placebo
- Cohort B (Experimental): Each subjects in Cohort B will receive 2 single doses of PF-06291874 and 1 placebo dose in random order in Periods 1-3; in addition, 1 dose of PF-06291874 will be administered in Period 4 in the fed state.
  Interventions: Drug: PF-06291874 or Placebo

INTERVENTIONS:
Drug: PF-06291874 or placebo — PF-06291874 will be administered as an extemporaneously prepared suspension for all doses within the initially planned range of 3 mg to 100 mg. Correspondingly, placebo doses will be administered as suspension.
  Arms: Cohort A
Drug: PF-06291874 or Placebo — PF-06291874 will be administered as an extemporaneously prepared suspension for all doses within the initially planned range of 300 mg to 650 mg. Correspondingly, placebo doses will be administered as suspension.
  Arms: Cohort B

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability, pharmacokinetics, and pharmacodynamics of single oral doses of PF-06291874 in healthy volunteers.

DETAILED DESCRIPTION:
The primary purpose of this trial is to evaluate the safety and tolerability, pharmacokinetics, and pharmacodynamics of single oral doses of PF-06291874 in healthy volunteers. The trial was terminated on Jan 9, 2012, due to undesired pharmacokinetic properties. The decision to terminate the trial was not based on any safety or efficacy concerns.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non childbearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including clinically significant drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability data: number of subjects with adverse events and Laboratory Test Values of Potential Clinical Importance, Changes from baseline in pulse rate, blood pressure and Electrocardiogram (ECG) measurements over 48 hrs | 2 days/dose group
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] - Fasted 0, 0.5, 1,2,3,4,6,8,12,16,24,36 and 48 hrs | 2 days/dose group
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) - Fasted 0, 0.5, 1,2,3,4,6,8,12,16,24,36 and 48 hrs | 2 days/dose group
Maximum Observed Plasma Concentration (Cmax) fasted - 0, 0.5, 1,2,3,4,6,8,12,16,24,36 and 48 hrs | 2 days/dose group
Time to Reach Maximum Observed Plasma Concentration (Tmax) -fasted 0, 0.5, 1,2,3,4,6,8,12,16,24,36 and 48 hrs | 2 days/dose group
Plasma Decay Half-Life (t1/2) fasted 0, 0.5, 1,2,3,4,6,8,12,16,24,36 and 48 hrs | 2 days/dose group
Apparent Oral Clearance (CL/F) fed 0, 0.5, 1,2,3,4,6,8,12,16,24,36 and 48 hrs | 2 days/dose group
Apparent Volume of Distribution (V/F) fed 0, 0.5, 1,2,3,4,6,8,12,16,24,36 and 48 hrs | 2 days/dose group

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4801001&StudyName=A%20Single%20Dose%20Study%20Of%20PF-06291874%20In%20Healthy%20Adult%20Subjects